CLINICAL TRIAL: NCT05736107
Title: A Randomized, Placebo-Controlled, Phase 2b Study to Evaluate the Efficacy, Safety and Tolerability of CBL-514 Injection for Reducing Abdominal Subcutaneous Fat
Brief Title: A Study to Evaluate the Efficacy, Safety and Tolerability of CBL-514 Injection for Reducing Abdominal Subcutaneous Fat
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Caliway Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBL-0204
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Subcutaneous Fat
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CBL-514 Injection (Experimental): Participant will receive CBL-514 2 mg/cm² administered in 2.4 mL injections, up to 120 mL per treatment session at intervals of approximately 3 weeks for up to a maximum of 4 treatments.
  Interventions: Drug: CBL-514 Injection
- 0.9% Sodium Chloride (Placebo Comparator): Participant will receive 0.9% Sodium Chloride administered in 2.4 mL injections, up to 120 mL per treatment session at intervals of approximately 3 weeks for up to a maximum of 4 treatments.
  Interventions: Other: 0.9% Sodium Chloride

INTERVENTIONS:
Drug: CBL-514 Injection — Formulated as an injectable CBL-514 solution at a concentration of 5 mg/mL.
  Arms: CBL-514 Injection
Other: 0.9% Sodium Chloride — Sodium Chloride (0.9% NaCl) placebo for injection
  Arms: 0.9% Sodium Chloride

SUMMARY:
This is a randomized, placebo-controlled, Phase 2b study to evaluate the efficacy, safety, and tolerability of CBL-514 injection for reducing subcutaneous fat.

DETAILED DESCRIPTION:
A total of approximately 110 adult participants with moderate or severe abdominal fat as assessed by the Investigator via live evaluation using the Clinician-Reported Abdominal Fat Rating Scale (CR-AFRS) at Screening will be enrolled. Each participant will receive up to 4 treatments of allocated CBL-514 (2 mg/cm²) or placebo administered subcutaneously to the abdomen, once every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 years to 64 years old (at Screening), inclusive.
2. Body mass index (BMI) > 18.5 and < 30 kg/m2 and body weight ≥ 50 kg at Screening and Day 1.
3. Participant has abdominal fat graded by the Investigator as Grade 3 (moderate) or Grade 4 (severe) using the Clinician-Reported Abdominal Fat Rating Scale via live evaluation at Screening.
4. Participant has stable body weight (identified as ≤ 3 kg weight change per participant report) for at least 3 months before Screening and during the study.
5. Participant who has maintained a stable lifestyle (e.g., exercise, eating patterns, and smoking habit) per participant report for at least 3 months before Screening and during the study.
6. Voluntarily signs the Informed Consent Form (ICF) and, in the opinion of the Investigator or delegate, is physically and mentally capable of participating in the study, and willing to adhere to study procedures.

Exclusion Criteria:

1. Female participant of childbearing potential who is not willing to commit to an acceptable contraceptive regimen from the time of Screening and throughout study participation until 90 days after the last IP dose, or who is currently pregnant or lactating. Male participant who is not willing to commit to using of a condom and refraining from sperm donation from the time of the first dose of IP, throughout study participation until 90 days after the last IP dose.

   Note: Participants who are not of childbearing potential are not required to use contraception. Females not of childbearing potential are defined as those who have been surgically sterilized (hysterectomy or bilateral oophorectomy) or who are post-menopausal (defined as at least 50 years of age with greater than or equal to 12 months of amenorrhea with a follicle stimulating hormone (FSH) greater than 30 IU/L).
2. Participant diagnosed with coagulation disorders or who is receiving anticoagulant/antiplatelet therapy or medications or dietary supplements that impede coagulation or platelet aggregation.
3. Participant has hemoglobin A1c (HbA1c) greater than or equal to 9%, delayed wound healing, or poorly controlled diabetes defined as requiring a change in glucose control medications (other than day to day variations in insulin requirements) within the 6 months prior to Screening or for whom a change in glucose control medications is anticipated during the study, or any diabetic risks that, in the opinion of Investigator, make the individual an inappropriate candidate for the study.
4. Participant with active or prior history of malignancies within 5 years before Screening or currently being evaluated for a possible malignancy, with the exception of adequately treated basal cell carcinoma of skin and in situ squamous cell carcinoma of skin at Investigator's discretion.
5. Participant with a history of human immunodeficiency virus (HIV)-1 infection or participant with active HIV infection at Screening with positive HIV antigen/antibody (Ag/Ab) combo test.
6. Participant with a history of trypanophobia, the extreme fear of medical procedures involving injections or needles, or who experiences vasovagal syncope and faints at the sight of blood or a needle.
7. Participant with folding fat or skin on abdomen in standing position.
8. Participant with severe or very severe abdominal visceral fat assessed by the Investigator using the visceral fat scale.
9. Participant with ventral abdominal or umbilical hernia or previous repair of same.
10. Participant has abnormal skin or local skin conditions at the treatment area, which, in the opinion of Investigator, would increase risk to the participant or inhibit safety or efficacy evaluation, including but not limited to any of the following:

    1. Skin manifestations of a systemic disease,
    2. Any abnormality of the skin or soft tissues of the area to be treated, such as scars, striae, dyspigmentation, etc.,
    3. Asymmetrical fat on abdomen,
    4. Lipomatosis syndromes (familial lipomatosis, nevus lipomatosis, Dercum's disease, etc.),
    5. Skin laxity on abdomen,
    6. Sensory loss or dysesthesia in the area to be treated,
    7. Tattoo(s) on the front and/or lateral side of abdomen.
11. Participant who has undergone the following procedures:

    1. Previous surgery that caused scar tissues on the anticipated treatment area before Screening or during the study, with the exception of laparoscopic surgery and surgery that resulted in minimal scar tissue determined at Investigator's discretion,
    2. Liposuction or abdominoplasty to the region to be treated before Screening or during the study,
    3. Aesthetic procedure for body contouring or fat reduction, e.g., cryolipolysis, ultrasonic lipolysis, low level laser therapy, EMSculpt, lipolysis injection to the region to be treated within 12 months before Screening or during the study.
    4. Using medication that is delivered via subcutaneous injection at the treatment area within 4 weeks before Screening or during the study.
12. Participant is on prescription or OTC weight reduction medication, weight reduction programs, or use of any GLP-1 agonists (e.g., semaglutide, terzepatide, liraglutide, etc.) (oral or injectable) within 6 months before Screening or during the study.
13. Participant is undergoing chronic steroid or immunosuppressive therapy, with the exception of oral steroid inhalation indicated for asthma management or topical steroid application for skin conditions that are not directly applied to or indirectly affect the treatment area.
14. Requiring continual use of any medication that is known to strongly inhibit or induce CYP1A2 enzymes, sensitive CYP1A2 substrates or drugs with narrow therapeutic index during the study that, in the opinion of the Investigator, may affect the evaluation of the study product or place the participant at undue risk.

    Note: If a participant needs to use the above mentioned therapeutic agents during the study for any reason, these therapeutic agents should not be used at least for 2 days prior to dosing and until 1 day post-dose.
15. Unable to receive local anesthesia (e.g., history of hypersensitivity to lidocaine).
16. Participant with known allergies or sensitivities to the IP or its components, medical history of urticaria, any drug allergy, or seasonal allergy that presents with skin-related symptoms. Participant with food allergies can be enrolled at the discretion of Investigator.
17. Participant with liver cirrhosis, with inadequate liver function at Screening defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, total bilirubin (TBIL), or gamma-glutamyl transferase (GGT) greater than 3.0 × upper limit of normal (ULN), or with any hepatic medical condition that would interfere with assessment of safety or efficacy.
18. Participant with any renal impairment, defined as:

    1. serum creatinine greater than 1.5 × ULN and blood urea nitrogen (BUN) greater than 1.5 × ULN, or
    2. estimated glomerular filtration rate (eGFR) less than 90 mL/min/1.73 m2, or who is currently on dialysis.

    Note: Participant with an eGFR greater than or equal to 60 and less than 90 mL/min/1.73 m2 at Screening should be evaluated by the Investigator for pre-existing disease or associated dysfunction. If mild decrease in eGFR is deemed not clinically significant or not related to dysfunction by the Investigator, the participant will not be excluded unless the Investigator deems it necessary.
19. Participant with contraindications to MRI imaging.
20. Use of any investigational drug or device within 3 months prior to Screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2024-05-20 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Participants with at least 1-grade improvement reported by Investigator using the Clinician-Reported Abdominal Fat Rating Scale | From baseline to 12 weeks after the final treatment
  The scale is a 5-point ordinal scale to assess the abdominal fat level

SECONDARY OUTCOMES:
Participants with at least 1-grade improvement reported by Investigator using the Clinician-Reported Abdominal Fat Rating Scale | From baseline to 4 weeks and 8 weeks after the final treatment
  The scale is a 5-point ordinal scale to assess the abdominal fat level
Participants with at least 2-grade improvement reported by Investigator using the Clinician-Reported Abdominal Fat Rating Scale | From baseline to 4 weeks, 8 weeks and 12 weeks after the final treatment
  The scale is a 5-point ordinal scale to assess the abdominal fat level
Participants with at least 1-grade improvement reported by participant using the Patient-Reported Abdominal Fat Rating Scale | From baseline to 4 weeks, 8 weeks and 12 weeks after the final treatment
  The scale is a 5-point ordinal scale to assess the abdominal fat level
Change in subcutaneous fat compared to baseline | From baseline to 4 weeks and 12 weeks after the final treatment
  Measured by MRI

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sheu, Study Director — Caliway Biopharmaceuticals Co., Ltd.
Locations (1):
- Investigational site 1, Pflugerville, Texas, United States